CLINICAL TRIAL: NCT00515879
Title: D-cycloserine Enhancement of Exposure in Social Phobia
Brief Title: Effect of D-cycloserine Plus Cognitive Behavioral Therapy on People With Social Phobia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stefan G. Hofmann, Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH078308 (NIH); R01MH078308 (NIH); R01MH075889 (NIH)
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Social Anxiety Disorder
Keywords: Generalized subtype
MeSH Terms: conditions — Phobia, Social | interventions — Cycloserine; Cognitive Behavioral Therapy; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT plus d-cycloserine (Experimental): Participants will receive cognitive behavioral therapy plus D-cycloserine
  Interventions: Drug: D-cycloserine; Behavioral: Cognitive behavioral therapy (CBT)
- CBT plus placebo (Placebo Comparator): Participants will receive cognitive behavioral therapy plus pill placebo
  Interventions: Behavioral: Cognitive behavioral therapy (CBT); Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 50 mg
  Other Names: Seromycin
  Arms: CBT plus d-cycloserine
Behavioral: Cognitive behavioral therapy (CBT) — CBT sessions aim to help participants become more comfortable with social situations.
Drug: Placebo — Same dosage as active pill
  Other Names: Sugar pill
  Arms: CBT plus placebo

SUMMARY:
This study will assess the effectiveness of D-cycloserine combined with cognitive-behavior therapy in treating people with social anxiety disorder.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is among the most common psychiatric conditions and is associated with significant distress and dysfunction in social situations. Although treatment with cognitive-behavior therapy (CBT) is known to help remedy SAD, many patients do not respond to this treatment and most do not reach full recovery. In CBT, patients undergo repeated and prolonged exposure practices to feared social situations to learn better ways to deal with anxiety in these settings. Exposure therapy is based on animal models of extinction of conditioned fears, and recent animal research has identified some of the core pathways and neurotransmitters involved in fear extinction. D-cycloserine (DCS) is a drug that appears to facilitate learning and the process of extinction of conditioned fear in both animals and humans. This study will assess the effectiveness of DCS combined with CBT in treating people with SAD.

Participants in this double-blind study will be randomly assigned to an active or control group. All participants will attend 18 study visits at the Center for Anxiety and Related Disorders over a 9-month period. There will be 12 CBT sessions of 90 minutes each and 6 assessment visits. The CBT sessions will help participants to become more comfortable with social situations. During 5 of the CBT sessions, participants will receive a pill containing either DCS or sugar (placebo). Assessment visits will include interviews, self-report questionnaires, and laboratory tests. These visits will occur at Weeks 1, 7, and 12 during treatment and at Months 3, 6, and 9 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for generalized social anxiety disorder (GSAD)
* Total score of greater than or equal to 60 on the LSAS
* Physical examination, electrocardiogram, and laboratory findings without clinically significant abnormalities

Exclusion Criteria:

* Lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders, or obsessive-compulsive disorder
* Eating disorder within the 6 months prior to study entry
* History of organic brain syndrome, mental retardation, or other cognitive dysfunction
* Substance or alcohol abuse or dependence (other than nicotine) within the 6 months prior to study entry or inability to refrain from alcohol use during the acute period of study participation
* Post-traumatic stress disorder within 6 months prior to study entry; entry of patients with other mood or anxiety disorders will be permitted if the social anxiety disorder is judged to be the predominant disorder
* Suicidal thoughts
* Taking concurrent psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers) within 2 weeks of study entry
* Significant personality dysfunction
* Serious medical illness or instability for which hospitalization may be likely within the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan G. Hofmann, PhD, Principal Investigator — Boston University; Mark H. Pollack, MD, Principal Investigator — Massachusetts General Hospital; Jasper A. Smits, PhD, Study Director — Southern Methodist University
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hofmann SG, Pollack MH, Otto MW. Augmentation treatment of psychotherapy for anxiety disorders with D-cycloserine. CNS Drug Rev. 2006 Fall-Winter;12(3-4):208-17. doi: 10.1111/j.1527-3458.2006.00208.x. PMID 17227287
- [Background] Otto MW, Basden SL, Leyro TM, McHugh RK, Hofmann SG. Clinical perspectives on the combination of D-cycloserine and cognitive-behavioral therapy for the treatment of anxiety disorders. CNS Spectr. 2007 Jan;12(1):51-6, 59-61. doi: 10.1017/s1092852900020526. PMID 17192764
- [Background] Hofmann SG, Meuret AE, Smits JA, Simon NM, Pollack MH, Eisenmenger K, Shiekh M, Otto MW. Augmentation of exposure therapy with D-cycloserine for social anxiety disorder. Arch Gen Psychiatry. 2006 Mar;63(3):298-304. doi: 10.1001/archpsyc.63.3.298. PMID 16520435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective participants were recruited between September 2007 and June 2011 through referrals to the three study sites (Boston University [BU], Massachusetts General Hospital [MGH], and Southern Methodist University [SMU]), from other area clinical facilities and programs, and from advertisements.
Pre-assignment Details: Study participants underwent a two-step screening evaluation, consisting of 1) telephone screening, and 2) psychiatric assessment and medical history taking with physical examination.
Groups:
- D-cycloserine-augmented CBT: Participants will receive D-cycloserine augmented cognitive behavioral therapy
- Placebo-augmented CBT: Participants will receive placebo augmented cognitive behavioral therapy
Period: Overall Study
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Started | 87 | 82
Completed | 62 | 62
Not Completed | 25 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT | Total
Number analyzed (Participants) | 87 | 82 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 82 | 169
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (7.89) | 30.5 (8.9) | 32.55 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 30 | 74
  Male | 43 | 52 | 95
Region of Enrollment [Number; unit: participants]
  United States | 87 | 82 | 169

OUTCOME MEASURES:

1. Primary Outcome: Social Phobic Disorders Severity and Change Form
Description: Social Phobic Disorders Severity and Change Form (SPD-SC Form; Liebowitz et al., 1992) is an expansion and adaptation of the Clinical Global Impression Scale (CGI) by Guy (1976) to SAD. Similar to the original CGI scale, the SPD-SC Form is rated by an independent evaluator on a 7-point scale to indicate severity (1=normal/not ill; 2 = minimally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most severely ill) and improvement (1=very much improved; 2=much improved; . 3=minimally improved' 4 = no change; 5=nimimal deterioration; 6=severe deterioration; 7=very severe deterioration). The primary outcome measure is units of a scale ranging from 1 (very much improved) to 7 (very severe deterioration).
Time Frame: Measured at Months 3 (immediately after treatment)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Number analyzed (Participants) | 87 | 82
Units on a scale | 2.68 [2.38 to 2.98] | 2.95 [2.64 to 3.27]

2. Primary Outcome: Liebowitz Social Anxiety Scale (LSAS)
Description: The Liebowitz Social Anxiety Scale (LSAS; Liebowitz, 1987) is a 24-item scale that provides separate scores for fear and avoidance in social and performance situations; it is widely used in treatment studies of SAD. Total scores range from 0 (no anxiety) to 144 (maximum).
Time Frame: Measured at Months 3
Measure: Mean (95% Confidence Interval); unit: LSAS scores
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Number analyzed (Participants) | 87 | 82
LSAS scores | 39.19 [34.79 to 43.59] | 42.44 [37.94 to 47.03]

3. Secondary Outcome: Social Phobia and Anxiety Inventory
Description: The Social Phobia and Anxiety Inventory (SPAI; Turner, Beidel, Dancu, and Stanley, 1989) is a 45-item self-report measure on the frequency (0 = Never, 1 = Very Infrequent, 2 = Infrequent, 3 = Sometimes, 4 = Frequent, 5 = Very Frequent, 6 = Always) of one's experiences. The inventory includes 32 items assessing somatic, cognitive, and behavioral symptoms of social anxiety and 13 items assessing agoraphobia. The final score is calculated by subtracting the agoraphobia subscale total (max = 78; min = 0) from the social phobia subscale total (max = 192; min = 0). Thus, the final total scores range from 0-114, where higher final scores indicate higher social anxiety.
Time Frame: Measured at Months 3, 6, and 9 post-treatment
Population: The number of analyzed participants differs from the overall number analyzed due to participant dropout between treatment and subsequent follow up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Number analyzed (Participants) | 87 | 82
score on a scale
  3 Months: number analyzed (Participants) | 75 | 64
  3 Months | 71.08 (28.585) | 73.74 (30.311)
  6 Months: number analyzed (Participants) | 66 | 58
  6 Months | 69.64 (32.188) | 71.97 (30.566)
  9 Months: number analyzed (Participants) | 69 | 54
  9 Months | 67.67 (31.847) | 67.74 (33.289)

4. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Endicott et al., 1993) is a 16-item self-report measure that rates aspects of quality of life, including physical health, mood, activities of daily living, and overall life satisfaction. Responses are scored on a 5 point scale. The maximum score is 70 (high satisfaction) and the minimum is 14 (low satisfaction); scores are generally expressed as a percentage of maximum total score (0-100).
Time Frame: Measured at Months 3, 6, and 9 post-treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of maximum
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Number analyzed (Participants) | 87 | 82
percentage of maximum
  3 Months: number analyzed (Participants) | 76 | 66
  3 Months | 67.77 (14.075) | 67.44 (14.00)
  6 Months: number analyzed (Participants) | 68 | 60
  6 Months | 66.32 (16.066) | 67.44 (14.872)
  9 Months: number analyzed (Participants) | 67 | 54
  9 Months | 67.08 (16.063) | 69.58 (11.761)

5. Secondary Outcome: Liebowitz Self-Rated Disability Scale
Description: Liebowitz Self-Rated Disability Scale (Schneier et al., 1994) is an 11-item scale assessing impairment specific to social anxiety. Current (past 2 weeks) and most severe lifetime impairment due to social anxiety disorder are rated on a 0-3 scale of degree of limitation (0=problem does not limit me at all; 3=problem limits me severely). The maximum score is 44 (severe impairment) and the minimum is 0 (no impairment).
Time Frame: Measured at Months 3, 6, and 9 post-treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT Plus D-cycloserine | CBT Plus Placebo
Number analyzed (Participants) | 87 | 82
score on a scale
  3 Months: number analyzed (Participants) | 78 | 66
  3 Months | 15.6117 (7.25681) | 14.0303 (7.79688)
  6 Months: number analyzed (Participants) | 70 | 62
  6 Months | 15.5283 (7.03686) | 14.4977 (7.98470)
  9 Months: number analyzed (Participants) | 69 | 59
  9 Months | 15.3269 (7.72461) | 14.3130 (7.62630)

6. Secondary Outcome: Range of Impaired Functioning Tool
Description: The Range of Impaired Functioning Tool (LIFE-RIFT, Leon et al., 2000) is a clinician rated scale assessing functioning in four domains: work, interpersonal relationships, recreation, and global satisfaction. Each domain is scored 0-5 (0=not applicable, 1=no impairment, 2=slight impairment, 3=mild impairment, 4=moderate impairment, 5=severe impairment). The total score is the sum of each domain's score, with a maximum score of 20 (severe impairment) and a minimum score of 4 (no impairment).
Time Frame: Measured at Months 3, 6, and 9 post-treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Number analyzed (Participants) | 87 | 82
score on a scale
  3 Months: number analyzed (Participants) | 78 | 82
  3 Months | 8.5256 (2.780) | 8.6667 (2.80841)
  6 Months: number analyzed (Participants) | 70 | 82
  6 Months | 8.6143 (2.67730) | 8.5430 (2.82987)
  9 Months: number analyzed (Participants) | 69 | 82
  9 Months | 8.6232 (2.80284) | 7.7458 (2.43957)

ADVERSE EVENTS:
Arm/Group | D-cycloserine-augmented CBT | Placebo-augmented CBT
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/82
Other Adverse Events (participants affected / at risk) | 0/87 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No